CLINICAL TRIAL: NCT04029805
Title: Evaluation of the Effect of a Combination of a Plant Extract (BSL_EP044) and Lactobacillus BSL_PS6 on Glucidic Metabolism in Women Suffering From Polycystic Ovary Syndrome and High Insulin Levels
Brief Title: Evaluation of a Combination of a Plant Extract and a Probiotic on Glucidic Metabolism in Women With PCOS and High Insulin Levels
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P044
Record Dates: First submitted 2019-07-22; First posted 2019-07-23 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Ovarian Syndrome; Insulin Resistance
Keywords: Polycystic ovarian syndrome; Extract plant; Probiotics; Insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination of a Plant Extract and a Probiotic (Experimental): Volunteers will take twice at day for 12 weeks a capsule containing the combination of a plant extract (BSL_EP044) and Lactobacillus BSL_PS6
  Interventions: Combination Product: Combination of a plant extract (BSL_EP044) and Lactobacillus BSL_PS6
- Placebo (Placebo Comparator): Volunteers will take twice at day for 12 weeks a capsule containing maltodextrin.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Combination of a plant extract (BSL_EP044) and Lactobacillus BSL_PS6 — Each participant will consume 2 capsules daily, in the morning and at night without any restriction in the diet nor in their habits of life.
  Arms: Combination of a Plant Extract and a Probiotic
Combination Product: Placebo — Each participant will consume 2 capsules daily, in the morning and at night without any restriction in the diet nor in their habits of life.
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the effect of the combination of a plant extract (BSL_EP044) and Lactobacillus BSL_PS6 on parameters of the glucidic metabolism, anthropometric parameters, hormonal levels and the menstrual cycle in women with polycystic ovary syndrome and high insulin levels.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most prevalent endocrinopathy in women, affecting 4-15% of those who are of childbearing age. It is a complex and heterogeneous disease in which the gynecological disorder coexist with metabolic problems such as insulin resistance.

The beneficial effect of the extract plant BSL-EP044 on glycemic metabolism in women with PCOS is widely studied and demonstrated and Lactobacillus BSL_PS6 appears to exert a synergistic effect by supplementing the effect of BSL-EP044. The hypothesis of our study is that the addition of the probiotic strain Lactobacillus BSL_PS6 to extract plant BSL-EP044 treatment may improve the beneficial effect of this one on insulin resistance and other metabolic alterations related to PCOS.

The main objective of the present study is to evaluate the effect of the combination of a Plant Extract (BSL_EP044) and Lactobacillus BSL_PS6 on parameters related to glycemic metabolism in women with polycystic ovary syndrome and high insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with polycystic ovarian syndrome according to the Rotterdam criteria.
* HOMA values between 2.5 and 3.
* Body mass index of less than 35 kg/m2.
* Accept freely to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Women in treatment with oral antidiabetics.
* Being pregnant or intending to get pregnant.
* Be in fertility treatment.
* To suffer from other diseases that affect the hormonal response or that could interfere with the glucidic metabolism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Plasma insulin | 12 weeks
  Levels of plasma insulin
Plasma glucose | 12 weeks
  Levels of plasma glucose
HOMA | 12 weeks
  Insulin sensitivity

SECONDARY OUTCOMES:
Total testosterone | 12 weeks
  Total testosterone
Free testosterone | 12 weeks
  Free testosterone

OTHER OUTCOMES:
Weight | 12 weeks
  Weight variation throughout the study
BMI | 12 weeks
  Body mass index
Blood pressure | 12 weeks
  Systolic and diastolic pressure during the study
Ovarian cycle | 12 weeks
  Duration of the ovarian cycle

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás Mendoza, MD, PhD, Principal Investigator — Professor of Gynecology at the Faculty of Medicine of the University of Granada
Locations (1):
- Clinica Margen, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No